CLINICAL TRIAL: NCT02521506
Title: Clinical Efficacy of OneTouch® Verio™IQ Meter
Acronym: ECOVIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ECOVIQ
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verio Pattern Alert® activated (Experimental): In this cohort, the patients will monitoring the glucose levels with capillar glucometer and they have activated the software Verio Pattern Alert® that could predict the glucose trends.
  Interventions: Device: Verio Pattern Alert® activated
- Verio Pattern Alert® deactivated (Active Comparator): In this cohort, the patients will monitoring the glucose levels with capillar glucometer.
  Interventions: Device: Verio Pattern Alert® deactivated

INTERVENTIONS:
Device: Verio Pattern Alert® activated
  Arms: Verio Pattern Alert® activated
Device: Verio Pattern Alert® deactivated
  Arms: Verio Pattern Alert® deactivated

SUMMARY:
Diabetes mellitus is one of the most prevalent disease in the western world. The control of glucose levels has a big impact in the prevention of diabetes complications. The measure of glucose levels in capillary blood with glucometers is the gold standard to measure and control the glucose levels. Nowadays the glucometers become to more precise and sophisticated devices. One of the most notables advance is the inclusion of software that cam predicts glucose trends. This software has not be tested in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with diabetes mellitus 1 or 2
* Treatment with insulin regimen during at least 12 months
* Capability of performed 3 glucose measurement per day
* Levels of glycated hemoglobin (A1C) less than 10%

Exclusion Criteria:

* Patients diagnosed of mental disorders
* Patients included in structured therapeutic health 6 months before the inclusion
* Patients included in any clinical trial in the 4 months before the inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
number of hypoglycemic events | 20 months
  Glucose levels under 70 mg/dL with or without clinical manifestation

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Universitario Torrecárdenas, Almería, Almería
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga